CLINICAL TRIAL: NCT06327841
Title: The Plaque Reducing Efficacy of Oil Pulling With Sesame Oil. A Randomized-controlled Clinical Study
Brief Title: Plaque Reduction Sesame Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Christine Zürcher, Dr.med.dent., Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK 1117/2022
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Dental Plaque; Gingivitis; Oral Microbial Colonization
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Sesame Oil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sesame oil (Experimental): 8 weeks oil pulling with sesame oil 15ml 15min every morning
  Interventions: Other: sesame oil
- distilled water (Other): 8 weeks rinsing with distilled water 15ml 15min every morning
  Interventions: Other: distilled water

INTERVENTIONS:
Other: sesame oil — 15min of oil pulling with 15ml sesame oil for 8 weeks
  Arms: sesame oil
Other: distilled water — 15min rinsing with 15ml distilled water for 8 weeks
  Arms: distilled water

SUMMARY:
The goal of this clinical trials to learn about potential additives in reducing dental plaque. The main questions it aims to answer is:

• is there a difference in the plaque reducing effect of oil pulling with sesame oil compared to rinsing with distilled water? Participants will rinse with 15 ml of their allocated liquid for 15 min every morning for 8 weeks.

Researchers will compare sesame oil against distilled water to see if there is a difference in the plaque reducing effect.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* contractual capability
* the presence of ≥ 10 teeth,
* community periodontal index of treatment needs (CPITN) grade 1 or 2

Exclusion Criteria:

* missing consent
* community periodontal index of treatment needs (CPITN) grade 0, 3 or 4
* pregnancy or breastfeeding
* systemic diseases or conditions that are associated with an increased risk of infection or necessitate concomitant antibiotic therapy with dental treatment
* mental and behavioral disorders that impede (verbal) communication
* allergy against sesame(oil)
* intake of antibiotics 6 months prior to or during study duration
* intake of medication potentially influencing gingival inflammation or bleeding (e.g. anticoagulants, cortisone)
* infectious diseases (e.g. HIV, hepatitis B or C)
* fixed orthodontic appliances
* ongoing oil pulling or mouth rinsing
* adult guardianship
* insufficient nasal breathing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Rustogi Modified Navy Plaque Index (RMNPI) | first follow up after 4 weeks, full study duration 8 weeks

SECONDARY OUTCOMES:
Gingival Index (GI) | first follow up after 4 weeks, full study duration 8 weeks
microbial analysis | first follow up after 4 weeks, full study duration 8 weeks
Oral Health Impact Profile (OHIP) | first follow up after 4 weeks, full study duration 8 weeks
Interview halitosis, xerostomia | first follow up after 4 weeks, full study duration 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ines Kapferer-Seebacher, Study Chair — Medical University Innsbruck; Markus Nagl, Study Chair — Medical University Innsbruck
Locations (1):
- Medical University, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zurcher C, Vukoje K, Kleiner EM, Kuster SM, Jager-Larcher LK, Heller I, Eick S, Nagl M, Kapferer-Seebacher I. The plaque reducing efficacy of oil pulling with sesame oil: a randomized-controlled clinical study. Clin Oral Investig. 2025 Jan 9;29(1):53. doi: 10.1007/s00784-024-06134-y. PMID 39786483